CLINICAL TRIAL: NCT02565030
Title: Chronic Thrombo-embolic Pulmonary Hypertension: Classification and Long Term Outcome
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH18804
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Idiopathic Pulmonary Arterial Hypertension
Keywords: Chronic thromboembolic Pulmonary Hypertension; Distal Chronic thromboembolic Pulmonary Hypertension; Proximal Chronic thromboembolic Pulmonary Hypertension; Operable disease; In-operable disease; Pulmonary Endarterectomy; PH specific targeted therapy; Phosphodiesterase type 5 Inhibitors; Endothelin Receptor Antagonist; Prostacyclin analogues; Soluble Guanylate cyclase stimulator; Sildenafil; Tadalafil; Bosentan; Ambrisentan; Macitentan; Iloprost; Riociguat; Idiopathic Pulmonary Arterial Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CTEPH surgical disease, operated: Patients with proximal CTEPH who have undergone Pulmonary Endarterectomy (PEA) surgery
- CTEPH surgical disease, not operated: Patients with proximal CTEPH with operable distribution of disease& have not undergone PEA surgery due to the following reasons:
  1. Multiple co-morbidities
  2. Patients choice
  3. Mild disease /symptoms
  4. Awaiting Surgery
- CTEPH non surgical: Patients with distal CTEPH with inoperable distribution of disease inaccessable to surgery.
- IPAH: Patients with IPAH as per European Society of Cardiology(ESC) criteria

SUMMARY:
This study will help to provide more up to date prognostic data on the natural history of untreated proximal CTEPH which will be helpful in discussions regarding surgical versus medical treatment and by exploring the similarities and differences between distal CTEPH and IPAH the investigators hope to get insights into disease mechanisms in patients with distal CTEPH.

DETAILED DESCRIPTION:
Chronic thrombo-embolic pulmonary hypertension (CTEPH) is thought to represent the consequence of failure of thrombus resolution after the establishment of thrombosis within the elastic pulmonary arteries. Thrombotic material becomes fibrosed, with occlusive vascular remodeling and the development of a secondary small vessel arteriopathy, termed the two-compartment model. This results in an increase in pressure and vascular resistance in the pulmonary vasculature and leads eventually to right heart failure.

It has been demonstrated that 2 year survival for CTEPH patients with mean pulmonary arterial pressure(mPAP) >50 mm Hg was only 20%, however, preliminary data from Sheffield Teaching Hospitals suggest that survival is significantly better than this. Until recently surgery was the only treatment for CTEPH in selected patients. Studies have shown the 10 year survival in patients with CTEPH after PEA surgery was 74%. More recently, for patients with inoperable CTEPH, drug therapy has been shown to improve exercise capacity. Despite recent publications the natural history and mechanisms underlying CTEPH are poorly understood.

The main area of research focus in this study will be improving understanding of the natural history of chronic thromboembolic pulmonary hypertension. The purpose of this research protocol is to conduct a retrospective review of patients with CTEPH diagnosed at the Sheffield Centre between 2001 and 2014 to understand more about the natural history of disease including prognostic indicators. The Sheffield Service has one of the largest cohorts of CTEPH in the world (>650 diagnosed cases since 2001). Approximately half of these patients undergo curative surgery with pulmonary endarterectomy. However, a significant proportion of patients with operable disease decline surgery and a significant proportion of patients have disease that is too distal for surgery, so called distal CTEPH. There is a relative paucity of data on i) the natural history of this disease, ii) an understanding of the relative contribution of obstruction and distal vasculopathy to elevations in pulmonary vascular resistance iii) the effects of distal CTEPH on right ventricular function and iv) how distal CTEPH differs from idiopathic pulmonary arterial hypertension (IPAH).

The second part of this study will focus on understanding disease mechanisms utilising MR imaging techniques and using the Sheffield PH Biobank resource to understand differences in the IPAH and distal CTEPH cohorts. The Sheffield PH Biobank has samples and detailed phenotypic data on over 400 treatment naïve patients with all forms of pulmonary hypertension with serial sampling and long term follow up providing a unique resource to make detailed comparisons across all forms of pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the diagnosis of chronic thromboembolic pulmonary hypertension and Idiopathic pulmonary arterial hypertension (as per the European Society of Cardiology guidelines) who presented to Sheffield Pulmonary Vascular Disease Unit at the Royal Hallamshire Hospital between 1st Jan 2001 and 1st Dec 2014.

Exclusion Criteria:

* Patients with Pulmonary Hypertension who have other causes of pulmonary hypertension in addition to chronic thromboembolic pulmonary hypertension and Idiopathic pulmonary arterial hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to Sheffield Pulmonary Vascular Disease Unit from the Midlands , North of England & Wales.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Death | Upto 176 months
  All patients with CTEPH or IPAH who have been documented as having died between 01/01/2001 and 01/09/2015

SECONDARY OUTCOMES:
Mean Pulmonary Arterial Pressure(mm of Hg) | Upto 176 months
  Measure of the final Mean Pulmonary Arterial Pressure with Right Heart Catheter studies in patients with CTEPH and IPAH reported between 01/01/2001 and 01/09/2015
Diffusion across the lung of Carbon Monoxide(mmol/min/KPa) | Upto 176 months
  Measure of final Diffusion across the lung of Carbon Monoxide in patients with CTEPH & IPAH reported between 01/01/2001 and of 01/09/2015
Emphasis 10 Quality Of Life Questionaire Score(0-50) | Upto 176 months
  Measure of the Emphasis 10 Quality of Life Questionaire Score in patients with CTEPH and IPAH in their final clinic visit reported between 01/01/2001 and 01/09//2015
Incremental Shuttle Walk Distance( in metres) | Upto 176 months
  The measure of the final Incremental Shuttle Walk Distance of patients with CTEPH and IPAH reported between 01/01/2015 and 01/09/2015
World Health Organization Functional Class(I-IV) | Upto 176 months
  Measure of the final World Health Organization Functional Class in patients with CTEPH and IPAH reported between 01/01/2001 and 01/09/2015
Right Ventricular Ejection Fraction(%) | Upto 176 months
  Measure of the final Right Ventricular Ejection Fraction with Cardiac Magnetic Resonance Imaging(MRI) in patients with CTEPH and IPAH reported between 01/01/2001 and 01/09/2015

CONTACTS AND LOCATIONS:
Overall Officials: Syed Quadery, MBBS, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; David Kiely, MD, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust; Wild Jim, PhD, Study Director — University Of Sheffield, School of Medicine; Andy Swift, MD, Study Director — University Of Sheffield , School Of Medicine
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Result] Riedel M, Stanek V, Widimsky J, Prerovsky I. Longterm follow-up of patients with pulmonary thromboembolism. Late prognosis and evolution of hemodynamic and respiratory data. Chest. 1982 Feb;81(2):151-8. doi: 10.1378/chest.81.2.151. PMID 7056079
- [Result] J Cannon, K Page, M Roots, A Ponnaberanam, C Tracy, D Taboada Buasso, K Sheares, C Ng, J Dunning, S Tsui, J Pepke-Zaba, D Jenkins.Outcome after Pulmonary Endarterectomy(PEA):Long term followup of UK National Cohort. Thorax 2013;68(Suppl 3):A25-A26.
- [Result] Hurdman J, Condliffe R, Elliot CA, Davies C, Hill C, Wild JM, Capener D, Sephton P, Hamilton N, Armstrong IJ, Billings C, Lawrie A, Sabroe I, Akil M, O'Toole L, Kiely DG. ASPIRE registry: assessing the Spectrum of Pulmonary hypertension Identified at a REferral centre. Eur Respir J. 2012 Apr;39(4):945-55. doi: 10.1183/09031936.00078411. Epub 2011 Sep 1. PMID 21885399
- [Result] Pepke-Zaba J, Delcroix M, Lang I, Mayer E, Jansa P, Ambroz D, Treacy C, D'Armini AM, Morsolini M, Snijder R, Bresser P, Torbicki A, Kristensen B, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Hamid AM, Jais X, Simonneau G. Chronic thromboembolic pulmonary hypertension (CTEPH): results from an international prospective registry. Circulation. 2011 Nov 1;124(18):1973-81. doi: 10.1161/CIRCULATIONAHA.110.015008. Epub 2011 Oct 3. PMID 21969018
- [Result] Condliffe R, Kiely DG, Gibbs JS, Corris PA, Peacock AJ, Jenkins DP, Goldsmith K, Coghlan JG, Pepke-Zaba J. Prognostic and aetiological factors in chronic thromboembolic pulmonary hypertension. Eur Respir J. 2009 Feb;33(2):332-8. doi: 10.1183/09031936.00092008. Epub 2008 Oct 1. PMID 18829679
- [Derived] Shahin Y, Alabed S, Alkhanfar D, Tschirren J, Rothman AMK, Condliffe R, Wild JM, Kiely DG, Swift AJ. Quantitative CT Evaluation of Small Pulmonary Vessels Has Functional and Prognostic Value in Pulmonary Hypertension. Radiology. 2022 Nov;305(2):431-440. doi: 10.1148/radiol.210482. Epub 2022 Jul 12. PMID 35819325
- [Derived] Quadery SR, Swift AJ, Billings CG, Thompson AAR, Elliot CA, Hurdman J, Charalampopoulos A, Sabroe I, Armstrong IJ, Hamilton N, Sephton P, Garrad S, Pepke-Zaba J, Jenkins DP, Screaton N, Rothman AM, Lawrie A, Cleveland T, Thomas S, Rajaram S, Hill C, Davies C, Johns CS, Wild JM, Condliffe R, Kiely DG. The impact of patient choice on survival in chronic thromboembolic pulmonary hypertension. Eur Respir J. 2018 Sep 16;52(3):1800589. doi: 10.1183/13993003.00589-2018. Print 2018 Sep. PMID 30002102